CLINICAL TRIAL: NCT04961866
Title: Effects of Parenteral Protein Concentrations in Critically Ill Patients in Icu (Comparative Study)
Brief Title: Effects of Parenteral Protein Concentrations in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Karim Naser Hasan, assisstant lecturer, Minia University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 308:10/2019
Record Dates: First submitted 2021-06-28; First posted 2021-07-14 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Hand Muscle Strain
Keywords: protein; parenteral; critical ill patient; ICU
MeSH Terms: interventions — Parenteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients received 1 g/ kg of protein
  Interventions: Dietary Supplement: parenteral protein 1 g/kg
- Group B (Active Comparator): patients received 2 g/ kg of protein
  Interventions: Dietary Supplement: Parenteral nutrition 2 g/kg

INTERVENTIONS:
Dietary Supplement: parenteral protein 1 g/kg — patients received 1 g/ kg of protein
  Arms: Group A
Dietary Supplement: Parenteral nutrition 2 g/kg — Patients received 2 g/ kg of protein
  Arms: Group B

SUMMARY:
Sixty patients who need Parenteral nutrition for more than 48h will be assigned into two groups .Group A (n=30) patient will receive 1g/kg/day protein and group B n=30) patient will receive 2g /kg/day. In both groups caloric requirement will be fixed at 25- 30 kcal /kg/d.

DETAILED DESCRIPTION:
In this study after obtaining approval from our hospital ethics committee, a written informed consent will be obtained from patient's next of kin.

Sixty patients who need PN for more than 48h will be assigned into two groups .Group A (n=30) patient will receive 1g/kg/day protein and group B n=30) patient will receive 2g /kg/day. In both groups caloric requirement will be fixed at 25- 30 kcal /kg/d.

Inclusion criteria:

Age: from 18 to 60 years Sex : male or female Predicted to be in icu ≥ 48 hs Predicted to have PN for> 48 hs.

Exclusion criteria:

Pregnant female Hepatic patients Renal patients Age <18 years

Technique of the study :

60 abdominal surgery/trauma ICU patients who have a contraindication or intolerance to enteral nutrition(EN),will be fed parenterally within 24-48 h from admission and divided according to the protein delivery into two groups.

Group A , those patients will receive parenteral proteins in a dose of 1 g/kg/day.

Group B, those patients will receive parenteral proteins in a dose of 2g/kg /day The nutrition will be delivered through a central line and using separate bottles technique ,because of the lack of a compounding unit and commercial bags in our hospital, After exclusion of the protein calories (will be given as 10%aa )the rest of energy requirement will be divided between carbohydrates (glucose25%)and lipids(SMOF20%) in a ratio of 60:40 Serum electrolytes, blood glucose, lipid profile and serum creatinine will be monitored and corrected regularly in every patient

The two groups will be compared as regarding the following :

hand grip strength Time of staying on Icu Time of staying in hospital Ultrasound biceps muscle thickness Nitrogen balances

ELIGIBILITY:
Inclusion Criteria:

* Age: from 18 to 70 years Sex : male or female Predicted to be in icu ≥ 48 hs Predicted to have PN for> 48 hs.

Exclusion Criteria:

- Hepatic patients Renal patients Age <18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
hand grip strength | 10 days
  hand grip strength using dynamometer

SECONDARY OUTCOMES:
ultrasound guided muscle thickness | 10 days
  us guided biceps and forearm muscle thickness
nitrogen balances | 10 days
  Measurements

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim A. Youssif, MD, Study Chair — Minia University
Locations (1):
- Karim Naser Hasan, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No